CLINICAL TRIAL: NCT03473626
Title: A Two-Period, Randomised, Crossover Study Designed to Evaluate the In Vivo Performance of a Modified Release Formulation of Alicaforsen in Healthy Male Subjects in the Fed and Fasted State
Brief Title: Phase 1 Food Effect Study for Alicaforsen Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atlantic Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ACH HV-AO-101
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: IBD
MeSH Terms: interventions — alicaforsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alicaforsen tablets (Experimental): Regimen A - Alicaforsen tablets with food
  Interventions: Drug: Alicaforsen
- alicaforsen tablets (Experimental): Regimen B - Alicaforsen tablets without food
  Interventions: Drug: Alicaforsen

INTERVENTIONS:
Drug: Alicaforsen — Alicaforsen tablet

SUMMARY:
Phase 1 study to compare the effect of food on alicaforsen tablet.

DETAILED DESCRIPTION:
A study on healthy male vounteers in a phase 1 unit. Alicaforsen tablets are gievn in a fed and fasted state

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer

Exclusion Criteria:

* Drugs of abuse
* Alcohol abuse

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 24 hours
  Area under the curve recovery of alicaforsen in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Chris Dunk, Study Director — Atlantic Pharmaceuticals
Locations (1):
- Phase 1 unit, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No